CLINICAL TRIAL: NCT05773859
Title: Induction of Neo-Antigen Specific Cytotoxic T Cells by Autologous Tumor Lysate-loaded Specialized Cross-Presenting Dendritic Cells in Epithelial Ovarian Cancer Patients Treated With Neoadjuvant Chemotherapy, the NEODOC Study
Brief Title: NEOadjuvant Dendritic Cell Vaccination for Ovarian Cancer
Acronym: NEODOC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEODOC
Record Dates: First submitted 2023-02-12; First posted 2023-03-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Epithelial Ovarian Cancer; Ovarian Carcinoma
Keywords: immunotherapy; dendritic cell vaccination; ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — CDC1 protein, S cerevisiae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XP-DC vaccinations (Experimental): Patients in this arm will receive XP-DC vaccination in addition to standard-of-care treatment.
  Interventions: Biological: XP-DC vaccinations

INTERVENTIONS:
Biological: XP-DC vaccinations — Autologous cross-presenting dendritic cells loaded with autologous tumor lysate and KLH
  Other Names: dendritic cell vaccine; cdc1

SUMMARY:
This goal of this single arm, single center, exploratory phase I/II clinical trial is to learn more about the immunological efficacy, safety and feasibility of an autologous tumor lysate-loaded autologous XP-DC (cDC1)-based vaccine in patients with ovarian cancer.

DETAILED DESCRIPTION:
Epithelial ovarian cancer (EOC) is the deadliest gynecological malignancy worldwide. Despite intensified treatment, 5-year overall survival rates only improved modestly over the last 20 years and remain low at around 30% for patients with advanced disease in the Netherlands. To this day, results from trials with the checkpoint inhibitors, that have revolutionized treatment in other cancer types, have been disappointing in EOC. Therefore, novel effective therapies are long awaited.

Recently, naturally circulating blood -derived dendritic cells (nDC) were shown to be potent in inducing cytotoxic immune responses and tumor regression in cancer patients. An even more specialized DC subset, referred to as cDC1 (conventional Dendritic Cells type 1) or XP-DC (specialized cross presenting DC) have shown their superiority in preclinical models. They are better at inducing cytotoxic T-cell responses against tumors after uptake of necrotic tumor cell material, a phenomenon called cross-presentation. This capability in cross-presentation makes XP-DC an ideal DC type in combination with tumor lysate-loading to induce immune responses against the scarce neoantigens present in EOC tumors.

The objective of this exploratory trial is to investigate the immunological efficacy as well as safety and feasibility of tumor-lysate loaded XP-DC in EOC patients undergoing (neo-)adjuvant chemotherapy. To this end 10 patients with stage III ovarian cancer will be included and offered a combined approach with DC vaccination in addition to standard-of-care chemotherapy and surgery. Extensive monitoring of the immune system throughout the course of the trial will be performed.

ELIGIBILITY:
Inclusion criteria

* Women over 18 years old with histologically confirmed primary epithelial ovarian cancer.
* Not amenable by primary debulking surgery and in need of neoadjuvant chemotherapy and interval debulking
* High-grade or low grade serous histology
* FIGO stage IIIb, IIIc, IVa or IVb if only lymph nodes ≤ 1cm above the diaphragm or in the groins
* Extensive abdominal spread of tumor
* WHO/ECOG performance status 0-1
* Neutrophils >1.5x 109/L, platelets >100x 109/L, hemoglobin >5,6 mmol/L (9.0 g/dl), estimated glomerular filtration rate > 45 ml/min/1.73m2 , AST/ALT <3 x ULN, serum bilirubin <1.5 x ULN (exception: Gilbert's syndrome is permitted)
* Expected adequacy of follow-up
* Postmenopausal or evidence of non-childbearing status or for women of childbearing potential: negative urine or serum pregnancy test, within 28 days of study treatment and confirmed prior to treatment on day 1. Postmenopausal is defined as:

  * Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments;
  * or surgical sterilisation (bilateral oophorectomy or hysterectomy).
* Informed consent

Exclusion criteria

* Recurrent ovarian cancer
* Histologies other than high grade serous ovarian cancer such as, but not restricted to, endometrioid, mucinous, clear cell or carcinosarcoma
* Unable and/or unwilling to undergo standard chemotherapy and interval debulking surgery
* FIGO stage I-IIb, IIIa or IVb with liver, spleen or lung metastases or lymph nodes above the diaphragm or in the groins > 1 cm
* History of any second malignancy, with the exception of adequately treated basal cell carcinoma, cervical cancer > 5 years ago or early stage breast cancer >10 years ago.
* Any serious clinical condition that may interfere with the safe administration of DC vaccinations
* Heart failure (NYHA class III/IV)
* Any uncontrolled co-morbidity, e.g. psychiatric or social conditions interfering which participation
* Unable to undergo a tumor biopsy
* Pregnancy or insufficient anti-conception if reproduction is still possible
* Active infection of Hepatitis B, C, HIV and syphilis
* Serious other active infections
* Known allergy to shell fish
* Auto immune disease (exception: vitiligo is permitted)
* History of organ allografts
* Chronic treatment with systemic immunosuppressive drugs (i.e. more than 10 mg prednisolone equivalent)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with an immunological response to XP-DC vaccination | At DTH skin test after the second vaccination (approximately study week 10)
  Immunologically responding patients are defined as:
  T cells isolated from vaccine challenged sites (DTH biopsies) that can be expanded and 1) express T cell receptors specific for the vaccine and 2) show effector functions measured by IFN-gamma secretion or cytolytic activity against tumor antigen expressing target cells.
  Immunologically non-responding patients are defined as:
  No T cells, or T cells isolated from DTH biopsies that cannot be expanded, or T cells that can be expanded but do not recognize tumor antigens, or can recognize tumor antigens but do not display T effector functions i.e. lysis of tumor cell targets or release of IFN-α.

SECONDARY OUTCOMES:
Safety as assessed by incidence of treatment-related adverse events | Throughout the treatment phase until 1 year of follow-up
  Toxicity will be assessed according to CTCAE version 4.03.
Feasibility of tumor lysate-loaded XP-DC vaccinations in patients with advanced EOC | Throughout the treatment phase until the last planned vaccination (approximately study week 23)
  Feasibility assessment will be based on reporting of:
  * the number of patients from whom a successful apheresis product can be obtained
  * the number of patients from whom (both quantitatively and qualitatively) sufficient tumor lysate can be obtained
  * the number of patients for whom a DC product can be manufactured that meets the prespecified criteria
  * the number of patients that has received the planned number of vaccinations.
Recurrence free survival (RFS) after 12 months | 1 year
  Percentage of patients alive without recurrence of disease after 12 months
Number of patients with complete pathological response | At time of debulking surgery (approximately study week 11)
  The number of patients with a complete pathological response

CONTACTS AND LOCATIONS:
Overall Officials: Nelleke Ottevanger, MD/PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All IPD underlying the results in the publication will be made available in an online data repository under restricted access.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available beginning no longer than 3 months after the publication with no end date

REFERENCES:
- [Derived] Koeneman B, Schreibelt G, Duiveman-de Boer T, Bos K, van Oorschot T, Pots J, Scharenborg N, de Boer A, Hins-de Bree S, de Haas N, de Goede A, Westdorp H, van Ham M, de Vries IJM, Ottevanger PB. NEOadjuvant Dendritic cell therapy added to first line standard of care in advanced epithelial Ovarian Cancer (NEODOC): protocol of a first-in-human, exploratory, single-centre phase I/II trial in the Netherlands. BMJ Open. 2025 Nov 9;15(11):e102184. doi: 10.1136/bmjopen-2025-102184. PMID 41213670